CLINICAL TRIAL: NCT04031755
Title: Comparison of the Pharmacodynamic and Tolerability Profiles of Minocycline Versus Placebo in Autism Spectrum Disorder: a Double-blind, Placebo-controlled, Crossover, Proof-of-concept Study
Brief Title: A Proof-of-Concept Study of Minocycline in Autism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIN001 - Minocycline in ASD
Record Dates: First submitted 2019-05-10; First posted 2019-07-24 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Autism; Autism Spectrum Disorder; Minocycline
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Minocycline versus Placebo (Experimental): Phase 1: 4 weeks of daily minocycline 100mg BID dosing
  2-week washout period
  Phase 2: 4 weeks of daily placebo dosing
  Interventions: Drug: Minocycline; Drug: Placebos
- Placebo versus Minocycline (Experimental): Phase 1: 4 weeks of daily placebo dosing
  2-week washout period
  Phase 2: 4 weeks of daily minocycline 100mg BID dosing
  Interventions: Drug: Minocycline; Drug: Placebos

INTERVENTIONS:
Drug: Minocycline — Minocycline 100 mg capsules or matching placebo will be prepared by the central investigational pharmacy at Cincinnati Children's Hospital Medical Center. Drug identity will be masked by over encapsulation of the study drug.
  Other Names: Minocin
Drug: Placebos — Minocycline 100 mg capsules or matching placebo will be prepared by the central investigational pharmacy at Cincinnati Children's Hospital Medical Center. Drug identity will be masked by over encapsulation of the study drug.

SUMMARY:
The purpose of the study is to determine if Minocycline shows initial evidence of efficacy, safety, and tolerability in youth with Autism Spectrum Disorder ages 12 to 22 years.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, crossover, proof-of-concept study that compares the pharmacodynamic and tolerability profiles of minocycline versus placebo in autism spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

1. 22 ≥ Age ≥12 years. Males and females included in study.
2. Diagnostic confirmation of Autism Spectrum Disorder as confirmed by gold standard clinical interview using DSM 5 criteria and administration of the Autism Diagnostic Observation Schedule-2, Module 3 or 4.
3. General good health as determined by physical exam, medical and psychiatric history and safety labs as defined by the PI or designee.
4. Male study participants who are sexually active with a female partner of childbearing potential must be surgically sterilized, practicing abstinence, or agree to use highly effective methods of birth control (defined below), and not rely on barrier methods and spermicide alone, from the time of screening until 1 week after final dose of study drug.
5. Female participants of childbearing potential may be included in the study provided they are practicing abstinence or are using a double barrier method from the time of screening until 1 week after the final dose of study drug. Participants using hormonal methods of birth control (oral, intravaginal, transdermal, injectable, or implantable) must be on a stable dose for at least three months prior to screening.
6. Whole brain absolute cumulative gamma power (30 to 80 Hz) with median cut off at 2.5 (upward adjusted)

Exclusion Criteria:

1. Allergy or hypersensitivity to any of the tetracyclines antibiotics.
2. Inability to swallow study drug.
3. Concomitant use of scheduled anti-inflammatory drugs with the exception of as needed ibuprofen or acetaminophen use.
4. Unstable dosing of any mood, anxiety or behavior medications in the 5 half-lives prior to Phase 1 baseline visit.
5. Concomitant use of scheduled benzodiazepines, baclofen, gabapentin, pregabalin, or supplements with impact on the GABA system.
6. Concomitant daily use of antacids
7. Concomitant use of oral acne medications (isotretinoin), not including lotions or creams applied to the skin
8. Concomitant use of any cannabinoid or related product.
9. Unstable seizure disorder as defined by any seizure in the 6 months prior to baseline visit and/or a change in any anti-convulsant drug dosing in the 60 days prior to study screen.
10. Abnormal baseline safety lab assessments including, but not limited to ALT or AST greater than 1.5x the upper limit of normal, elevated ANA, total bilirubin or creatinine greater than 1x the upper limit of normal, other clinically relevant lab abnormality, or abnormality in ECG, HR or BP at screening as determined by the investigator or designee.
11. History of autoimmune disorder
12. History of or current abuse of drugs or alcohol including prescription medication.
13. Women who are pregnant (i.e. have a positive pregnancy test), intending to become pregnant, breast feeding, or women of child-bearing potential who are unwilling to use contraception as required in the study inclusion criteria or maintain abstinence during the course of the study
14. Inability to attend scheduled study visits, plans for family relocation during the study, or any other criteria that the investigator may determine to be associated with inability to complete the study

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Subject weight will be compared pre- and post-treatment in the drug versus placebo conditions | Through study completion, an average of 2 years
  Subject weight will be measured in kilograms
Aberrant Behavior will be evaluated pre- and post-treatment in the drug versus placebo conditions | Through study completion, an average of 2 years
  Aberrant behavior will be measured by the Aberrant Behavior Checklist total score
Incidence of liver toxicity will be evaluated in the pre- and post-treatment setting in the drug versus placebo conditions | Through study completion, an average of 2 years
  Liver toxicity will be defined as the development of an ALT or AST value greater than twice the upper limit of normal during a treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Craig Erickson, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Thompson Center for Autism & Neurodevelopmental Disorders - University of Missouri, Columbia, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Center for Autism and Developmental Disorders - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No